CLINICAL TRIAL: NCT06903572
Title: The Impact of Clinical Pharmacists Role in Transition of Care From Other Departments to Critical Care Units in Alexandria Main University Hospital.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Heba Shaker, Supervisor of clinical pharmacy units in ICU in Alexandria Main University Hospital, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0307050
Record Dates: First submitted 2025-03-25; First posted 2025-03-31 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-03

CONDITIONS: Intensive Care Admission

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients transmitted from other deprtments to to critical care department (Experimental)
  Interventions: Other: the clinical pharmacists interventions about medication related information during transition of care

INTERVENTIONS:
Other: the clinical pharmacists interventions about medication related information during transition of care — the intervention is the clinical pharmacists ' interventions regarding medication related information during transition of care .This includes reviewing medications regimen and treatment plan , documenting patients' drug history, drug related adverse events and detecting medication discrepancies.

SUMMARY:
Transition of care between hospital departments is an important step in patient care. Every patient may need to be transmitted either for case deterioration, improvement or interventions purposes. It includes patient transition from home to hospital, transition from one hospital to another, transition from one department to another in the same hospital, transition from hospital to home. This step has many patient safety risks due to health care teams' miscommunications, shifts handoffs and use of hard copies patients' profiles crowded with papers. So many pharmaceutical and health care organizations mentioned transition of care as one of patient and organizational related quality standards . All health care team members, including clinical pharmacists, have important roles to be played. Clinical pharmacists' services differ according to the setting at which patients are presented in.

They include medication reconciliation, resolution of medications discrepancies and medication related problems, interprofessional collaboration and communication, recommendations to patients and care givers and their engagement in the therapeutic plan and post discharge follow up .

ACCP structured task force recommendations for quality measures and associated metrics according to Avedis Donabedian's model of health care quality. Process metrics involve measuring the proportion of patients receiving transition of care services and calculating the total number of medication discrepancies and medication therapy problems and their distribution, overall and by type. Outcome measures include rates of unplanned 30 days, all cause hospital readmissions, total hospital length of stay, completion rates of first planned follow-up contact within prespecified time intervals as completion of post discharge telephone interview within 72 hours and completion rates of pharmacist-referred visits for preventive medicine or other medication-related concerns.

In this study ,the investigators will focus on clinical pharmacist services within transition in the same hospital from other department to critical care units. the investigatorswill select to measure the most important and applicable outcomes regarding this step of transition.

ELIGIBILITY:
Inclusion Criteria:All patients transmitted from any department in the hospital to critical care units.

-

Exclusion Criteria:Patients transmitted from other hospitals.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
the number of prescriptions with accurate medication use information after transition of patients to critical care reviewed by clinical pharmacists compared to that reviewed by critical care physicians. | 2 months
  the number of prescriptions with accurate medication use information (ex: dose, indication, duration, medications should be stopped or added, medications should be monitored) , after transition of patients to critical care reviewed by clinical pharmacists compared to that reviewed by critical care physicians.

SECONDARY OUTCOMES:
the total number of detected medication discrepancies and drug related problems and the number in each category | 2 months
  Counting the detected medication discrepancies and drug related problems and categorizing them by type (ex: inaccurate dose, inaccurate route of administration, duplication and unnecessary medications).

OTHER OUTCOMES:
length of patients stay in ICU | 2 months
  length of patients stay in ICU (total number of days)
mortality rate in patients whom benefited from clinical pharmacists service | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Main University Hospital, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided